# Studio prospettico osservazionale sull'incidenza di infezioni fungine invasive in pazienti affetti da leucemia linfoblastica acuta Ph-negativa

#### Studio SEIFEM ALL-IFI 2022

## **SEIFEM Writing Committee**

Chiara Cattaneo (UO di Ematologia, Spedali Civili di Brescia - CENTRO COORDINATORE)

Francesco Marchesi (UO Ematologia, Istituto Nazionale Tumori Regina Elena, Roma)

Irene Terrenato (UOSD Clinical Trial Center e Biostatistica e Bioinformatica, Istituto Nazionale Tumori Regina Elena, Roma)

Alessandro Busca (Chairman of the SEIFEM group)

Livio Pagano (President of the SEIFEM group)

## Introduzione

Le infezioni fungine invasive (IFI) sono una patologia opportunistica grave che si sviluppa tipicamente nel paziente immunocompromesso. Storicamente, in ambito ematologico, il setting della leucemia mieloide acuta (LMA) e quello del trapianto allogenico (alloSCT) sono stati considerati tra le condizioni maggiormente favorenti l'insorgenza di queste complicanze (1). Recentemente, tuttavia, sono stati pubblicati dati che evidenziano un incremento dell'incidenza delle IFI nei pazienti affetti da leucemia linfoblastica acuta (LLA), in particolare nelle Ph neg, rispetto ai dati storici, che collocavano la LLA come una condizione di rischio inferiore rispetto alla LMA e all'alloSCT (1, 2). In particolare, l'utilizzo di protocolli con schemi intensivi "pediatric-like" nella popolazione adulta e l'età avanzata sembrano essere una condizione di rischio per lo sviluppo delle complicanze infettive, con incidenze di IFI proven/probable che superano il 10% (3-5). Anche per le LLA Ph-neg, come per le LMA, l'incidenza è massima soprattutto in induzione (6), mentre per le LLA Ph-pos, dove gli schemi di chemioterapia sono più attenuati in quanto associati agli inibitori di tirosin-kinasi, l'incidenza di complicanze infettive è minore (2). Questi dati, tuttavia, sono estrapolati da studi clinici o si riferiscono a casistiche retrospettive, mentre gli studi prospettici sono carenti in questo ambito.

Il problema delle IFI nelle LLA rimane dunque una questione irrisolta, probabilmente anche perché, ad oggi, non è stata identificata una profilassi efficace utilizzabile in questo setting. L'utilizzo degli azoli, infatti, è controindicato per le interazioni farmacologiche con gli alcaloidi della vinca, mentre L-AmB non ha dimostrato una superiorità significativa rispetto al placebo nello studio AmbiGuard (7) e anche in uno studio retrospettivo di coorte (8). L'utilizzo di echinocandine rimane pure controverso, vista anche l'esiguità dei dati a disposizione nelle LLA (6, 8).

Per tali motivi, si ritiene fondamentale acquisire dati di *real life* circa il problema IFI nelle LLA Ph neg, mediante uno studio prospettico multicentrico, che possa rilevare l'incidenza delle IFI durante l'induzione.

## **Obiettivo primario**

Documentare la comparsa di infezioni fungine durante le prime fasi della chemioterapia (dall'esordio al TP2, ovvero alla 16 settimana) nei pazienti adulti affetti da LLA Ph-neg

#### Obiettivi secondari

- Documentare la comparsa di IFI in relazione alla profilassi antifungina adottata
- Documentare la comparsa di IFI in relazione all'età dei pazienti
- Documentare la comparsa di IFI in relazione alla durata della neutropenia
- Documentare la comparsa di IFI in relazione al tipo di trattamento steroideo adottato (desametazone sì vs no)
- Documentare eventuali ritardi nell'inizio della chemioterapia di consolidamento nei pazienti con LLA affetti da IFI
- Documentare l'outcome dei pazienti con LLA affetti da IFI

## Disegno dello studio

Lo studio è di tipo prospettico e osservazionale, multicentrico, di real-life che coinvolgerà XX centri afferenti al gruppo SEIFEM. Verranno arruolati tutti i pazienti affetti da LLA Ph-neg di età maggiore o uguale a 18 anni trattati con chemioterapia intensiva a partire dall'01.06.22 per la durata

di 18 mesi (+12 mesi di follow-up). La diagnosi di IFI verrà definita secondo i criteri EORTC 2019 (9). Le informazioni cliniche verranno raccolte in CRF cartacee, redatte in forma anonima.

L'incidenza di IFI e di aspergillosi polmonare durante la chemioterapia di induzione verrà messa in relazione alle seguenti variabili:

- Età
- Sesso
- Tipo di profilassi AF effettuata
- Classificazione del rischio LLA secondo i criteri ESMO 2016 (10)
- Dose di desametazone somministrata
- Durata della neutropenia
- Risposta ematologica e molecolare

#### Criteri di inclusione

- Pazienti affetti da LLA B Ph-neg o T all'esordio
- Età > 18 aa al momento dello studio
- Firma consenso informato

## Criteri di esclusione

- Pazienti affetti da LLA Ph-pos
- Pazienti affetti da LLA in recidiva
- Pazienti affetti da linfoma linfoblastico B/T

## **Endpoint primario**

Incidenza di IFI durante le prime fasi della chemioterapia (dall'esordio al TP2, ovvero alla 16 settimana) in pazienti affetti da LLA Ph-neg.

## **Endpoint secondari**

- Incidenza di IFI in pazienti affetti da LLA Ph-neg durante l'induzione in relazione alla profilassi antifungina adottata

- Incidenza di IFI in pazienti affetti da LLA Ph-neg durante l'induzione in relazione all'età
- Incidenza di IFI in pazienti affetti da LLA Ph-neg durante l'induzione in relazione alla durata della neutropenia
- Incidenza di IFI in pazienti affetti da LLA Ph-neg in relazione al tipo di trattamento steroideo adottato (desametazone sì vs no)
- Tempo mediano intercorso tra l'inizio effettivo della chemioterapia di consolidamento rispetto a quanto previsto dallo schema nei pazienti con LLA Ph-neg con IFI
- Tasso di mortalità dei pazienti in pazienti affetti da LLA Ph-neg con IFI

## Durata dello studio

Verranno arruolati tutti i pazienti eleggibili a partire dal 01.03.2022 per una durata di 18 mesi. Il tempo di follow-up dopo l'arruolamento sarà di 12 mesi.

#### Gestione dei dati

Tutti i dati saranno raccolti in forma anonima e a ciascun caso verrà assegnato un codice identificativo. I dati saranno conservati presso la S.C. di Ematologia dell'ASST-Spedali Civili di Brescia e saranno accessibili solamente ai soggetti coinvolti nello studio sopra citati.

#### **Statistica**

Lo studio proposto è un registro prospettico, multicentrico, osservazionale e di tipo clinico-epidemiologico. Prevede la partecipazione di 26 centri ematologici che dal 01.06.2022 tratteranno pazienti di età maggiore o uguale a 18 anni affetti da LLA Ph neg, per una durata di 18 mesi (+ 3 mesi di follow-up). La raccolta dati verrà effettuata tramite una CRF cartacea e opportunamente inseriti in un database elettronico, compilato con omissione di qualsiasi riferimento che possa permettere l'identificazione del paziente. Si chiederà il consenso informato all'uso dei dati a tutti i pazienti. La scheda raccolta-dati raccoglierà, per ogni paziente, informazioni relative sia alla patologia di base del paziente (tipo di diagnosi, numero di globuli bianchi all'esordio, caratteristiche biologicocitogenetiche, eventuali localizzazioni extramidollari), che relative all'infezione ed al suo decorso (profilassi antifungina ricevuta, tipo di infezione, gravità dell'infezione, trattamento ricevuto,

outcome clinico). La raccolta delle CRF consentirà di creare un ampio ed unico database multicentrico costruito con la partecipazione di tutti i centri ematologici che hanno trattato pazienti con le caratteristiche sopra-citate.

Una volta terminata la raccolta dati, si procederà all'analisi statistica finalizzata alla valutazione della distribuzione degli eventi infettivi fungini (IFI) ed all'identificazione dei parametri che influenzano significativamente l'insorgenza e l'outcome della complicanza infettiva.

## Dimensione campionaria

Il numero di pazienti arruolati si baserà sul numero di pazienti con LLA Ph negativa di età superiore o uguale a 18 anni che verranno sottoposti a chemioterapia di induzione presso i centri SEIFEM che aderiranno allo studio. Considerando il numero di centri che hanno dato adesione (26), il lasso temporale previsto per l'arruolamento (18 mesi) e la rarità della patologia in questione, si stima di arruolare complessivamente circa 150 pazienti. Basandoci su dati di letteratura che riportano un'incidenza di IFI durante l'induzione in pazienti con LLA Ph neg pari al 12% (4, 7), con una numerosità complessiva di 150 pazienti, una potenza statistica dell'80% e un livello di significatività del 5% (test binomiale a due code), ci aspettiamo un tasso di incidenza di IFI pari al 5.5%.

## Metodologia statistica

Il campione verrà presentato nelle sue caratteristiche cliniche e demografiche attraverso tecniche di statistica descrittiva. Le variabili quantitative verranno descritte con valori mediani e relativi range interquartili mentre quelle qualitative verranno presentate con frequenze assolute e percentuali. I potenziali fattori di rischio per l'evento infettivo verranno valutati tramite modelli di regressione logistica univariati e, per le variabili risultate statisticamente significative, verranno condotti modelli multivariati. Gli Odd Ratio stimati saranno accompagnati dai relativi intervalli di confidenza al 95% (95%IC) Un valore di p < 0.05 verrà considerato statisticamente significativo. L'analisi statistica sarà effettuata con software statistico (SPSS, versione 21.0). Lo studio non prevede alcuna spesa relativa alla raccolta dati o ad esami aggiuntivi. Tutti i dati raccolti afferiranno ad un centro coordinatore e saranno convogliati in un unico e omnicomprensivo database. Le reazioni avverse verranno segnalate analogamente a quanto previsto dalle norme in vigore per le segnalazioni spontanee (post-marketing).

## **Bibliografia**

- 1. Pagano L, Caira M, Candoni A, et al. The epidemiology of fungal infections in patients with hematologic malignancies: the SEIFEM-2004 study. Haematologica. 2006 Aug;91(8):1068-75.
- Pagano L, Busca A, Candoni A, et al. Risk stratification for invasive fungal infections in patients with hematological malignancies: SEIFEM recommendations. Blood Rev. 2017 Mar;31(2):17-29.
- 3. Doan TN, Kirkpatrick CM, Walker P, et al. Primary antifungal prophylaxis in adult patients with acute lymphoblastic leukaemia: a multicentre audit. J Antimicrob Chemother. 2016 Feb;71(2):497-505.
- 4. Gründahl M, Wacker B, Einsele H, Heinz WJ. Invasive fungal diseases in patients with new diagnosed acute lymphoblastic leukaemia. Mycoses. 2020 Oct;63(10):1101-1106.
- 5. Henden A, Morris K, Truloff N, et al. Incidence and outcomes of invasive fungal disease in adult patients with acute lymphoblastic leukemia treated with hyperfractionated cyclophosphamide, vincristine, doxorubicin and dexamethasone: implications for prophylaxis. Leuk Lymphoma. 2013 Jun;54(6):1329-31.
- 6. Cattaneo C, Gramegna D, Malagola M, et al. Invasive pulmonary aspergillosis in acute leukemia: a still frequent condition with a negative impact on the overall treatment outcome. Leuk Lymphoma. 2019 Dec;60(12):3044-3050.
- 7. Cornely OA, Leguay T, Maertens J, et al. Randomized comparison of liposomal amphotericin B versus placebo to prevent invasive mycoses in acute lymphoblastic leukaemia. J Antimicrob Chemother. 2017 Aug 1;72(8):2359-2367.
- 8. Batchelor R, Thomas C, Gardiner BJ, et al. When Azoles Cannot Be Used: The Clinical Effectiveness of Intermittent Liposomal Amphotericin Prophylaxis in Hematology Patients.

  Open Forum Infect Dis. 2021 Mar 8;8(7):ofab113.
- 9. Donnelly JP, Chen SC, Kauffman CA, et al. Revision and Update of the Consensus Definitions of Invasive Fungal Disease From the European Organization for Research and Treatment of Cancer and the Mycoses Study Group Education and Research Consortium. Clin Infect Dis. 2020 Sep 12;71(6):1367-1376.

Hoelzer D, Bassan R, Dombret H, et al. Acute lymphoblastic leukaemia in adult patients:
 ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016
 Sep;27(suppl 5):v69-v82.

11.

#### 12. SCHEDA INFORMATIVA

13.

- 14. Gentile Signora/e,
- 15. Lei è stato invitato a partecipare ad uno studio prospettico dal titolo: Studio prospettico osservazionale sull'incidenza di infezioni fungine invasive in pazienti affetti da leucemia linfoblastica acuta Ph-negativa". Questa ricerca è a carattere multicentrico, vale a dire sono interessati diversi Ospedali e Centri di Cura in Italia.
- 16. Per svolgere tale ricerca abbiamo bisogno della collaborazione e disponibilità di persone che, come Lei, sono affette da leucemia linfoblastica acuta Ph-negativa e ricevono un trattamento con chemioterapia. Comunque, prima che Lei prenda la decisione di accettare o rifiutare di partecipare, La preghiamo di leggere con attenzione, prendendo tutto il tempo che Le necessita, queste pagine e di chiedere chiarimenti al suo medico dello studio qualora non comprendesse o avesse bisogno di ulteriori precisazioni. Inoltre, qualora lo desiderasse, prima di decidere, può chiedere un parere ai suoi familiari o ad un suo medico di fiducia.

#### 17. CHE COSA SI PROPONE LO STUDIO

18. Si tratta di uno studio prospettico, multicentrico, osservazionale. Questo studio prevede l'arruolamento di tutti i pazienti affetti da a partire dall'1 Giugno 2022 per la durata di 18 mesi. Nello studio saranno arruolati i pazienti con leucemia linfoblastica acuta Ph-negativa in trattamento con chemioterapia. Lo studio ha come obiettivo generale quello di identificare, mediante indagini di tipo epidemiologico e clinico-laboratoristiche, l'insorgenza di infezioni fungine. Lei sarà seguito nelle diverse fasi di terapia e saranno raccolti i suoi dati anamnestici, clinici e di laboratorio attraverso la compilazione di un database da parte del suo medico dello studio. Verranno valutati i dati riguardanti l'infezione, il trattamento ed il decorso dell'infezione.

## 19. QUALI SONO I BENEFICI CHE POTRÀ RICEVERE PARTECIPANDO ALLO STUDIO

20. Dalla partecipazione a questo studio non sono prevedibili benefici diretti per Lei. La Sua partecipazione allo studio, però ci consentirà di acquisire maggiori conoscenze scientifiche sull'incidenza di infezioni fungine in pazienti affetti da leucemia linfoblastica acuta Ph-negativa che ricevono un trattamento con chemioterapia, informazione che consentirà in futuro di migliorare gli approcci terapeutici per i pazienti che saranno affetti dalla Sua stessa patologia.

#### 21. QUALI SONO I RISCHI DERIVANTI DALLA PARTECIPAZIONE ALLO STUDIO

22. La partecipazione allo studio non comporterà per lei alcun rischio, in quanto non è prevista la somministrazione di alcun farmaco, né l'esecuzione di indagini, ma la sola raccolta dei suoi dati anamnestici, clinici e di laboratorio attraverso la compilazione di alcune schede da parte del suo medico dello studio. Qualora divengano disponibili dati che possano influenzare la Sua volontà di continuare a partecipare allo studio, sarà tempestivamente informato/a.

# 23. INDAGINI A CUI SARÀ SOTTOPOSTO/A DURANTE LO STUDIO

**24.** Lo studio non prevede l'effettuazione di indagini di controllo al di fuori di quelle routinariamente eseguite nel caso della sua patologia.

#### 25. COSA SUCCEDE SE DECIDE DI NON PARTECIPARE ALLO STUDIO

26. Lei è libero/a di non partecipare allo studio. In questo caso riceverà, comunque, tutte le terapie standard previste per la Sua patologia, senza alcuna penalizzazione, ed i medici dello studio continueranno a seguirla comunque con la dovuta attenzione assistenziale.

#### 27. INTERRUZIONE DELLO STUDIO

28. La Sua adesione a questo programma di ricerca è completamente volontaria e Lei si potrà ritirare dallo studio in qualsiasi momento.

#### 29. INFORMAZIONI CIRCA I RISULTATI DELLO STUDIO

30. Se Lei lo richiederà, alla fine dello studio potranno esserLe comunicati i risultati dello studio in generale.

## 31. ULTERIORI INFORMAZIONI

- 32. Per ulteriori informazioni e comunicazioni durante lo studio sarà a disposizione il seguente personale: ...............
- 33. Deve impegnarsi a comunicare al suo medico di fiducia e a tutti gli altri medici con i quali si ponga in cura, il suo arruolamento nello studio osservazionale. Deve inoltre autorizzare il medico dello studio a contattare gli altri suoi medici curanti.
- 34. Il protocollo dello studio che Le è stato proposto è stato redatto in conformità alle Norme di Buona Pratica Clinica della Unione Europea e alla revisione corrente delle Dichiarazione di Helsinki ed è stato approvato dal Comitato Etico di questa struttura.
- 35. Le comunichiamo che i suoi dati personali saranno trattati in ottemperanza al D.Lgs. 30/06/2003 n.196 e Delibera del Garante 24/07/08 n.52 (Codice in materia di protezione dei dati personali).

| 36. | DICHIARAZIONE D | I CONSENSO |
|---|---|---|
| 37. | | |
| 38. | | |
| 39.<br>40. | | |
| | ichiaro di aver ricevuto dal Dottor <sup>1</sup> | |
| 42. | esaurienti spiegaz | oni in merito alla richiesta di partecipazione allo studio osservazionale in |
| | oggetto, secondo | quanto riportato nella scheda informativa qui allegata, copia della quale mi è |
| stata prima d'ora consegnata. | | |
| 43. | Dichiaro altresì di | aver potuto discutere tali spiegazioni, di porre tutte le domande che ho ritenuto |
| | necessarie e di ave | er ricevuto risposte soddisfacenti, come pure di aver avuto la possibilità di |
| | informarmi in mer | nformarmi in merito ai particolari dello studio con persona di mia fiducia. |
| 44. | unicare al mio medico di fiducia, e a tutti gli altri medici con i quali mi pongo in | |
| | cura, il mio arruola | amento nello studio osservazionale |
| 45. Autorizzo, il medico dello studio a contattare gli altri miei medici curanti. | | |
| 46. | Accetto liberamen | te di partecipare allo studio, avendo capito completamente il significato della |
| | richiesta e avendo compreso i rischi e i benefici che sono implicati. | |
| 47. | ato, inoltre del mio diritto ad avere libero accesso alla documentazione relativa | |
| | alla sorveglianza e | za ed alla valutazione espressa dal Comitato Etico e ad essere informato sui risultati |
| | dello studio in gen | erale. |
| 48. | Sono consapevole che i miei dati personali saranno trattati in ottemperanza al D.Lgs. 30/06/2003 | |
| | n.196 e Delibera d | el Garante 24/07/08 n.52 (Codice in materia di protezione dei dati personali). |
| 49. | | |
| | | <del></del> |
| Data | | Firma del medico che ha informato il paziente |
| Data | | Firma del paziente |

 $<sup>^{\</sup>rm 1}$  Indicare il nome del medico che ha informato il paziente sulla sperimentazione proposta.

| 50. |
|---|
| 51. [Nel caso il paziente non possa leggere e/o firmare]² |
| 52. |
| 53. lo sottoscritto: |
| 54. testimonio che il Dottor |
| 55. ha esaurientemente spiegato al Sig |
| 56. le caratteristiche dello studio in oggetto, secondo quanto riportato nella scheda informativa qu |
| allegata, e che lo stesso, avendo avuto la possibilità di fare tutte le domande che ha ritenuto |
| necessarie, ha accettato liberamente di aderire allo studio. |
| 57. |
| 58. |

| Data | Firma del testimone indipendente |
|------|----------------------------------|
| 59. | |
| 60. | |
| 61. | |
| 62. | |
| 63. | |
| 64. | |
| 65. | |
| 66. | |
| 67. | |
| 68. | |
| 69. | |
| 70. | |
| 71. | |
| 72. | |
| 73. | |
| 74. | |
| 75. | |
| 76. | |

<sup>&</sup>lt;sup>2</sup> Se il paziente non è in grado di leggere o di firmare, un testimone indipendente dallo sperimentatore e dallo sponsor deve essere presente durante l'intera discussione relativa al consenso informato. Il testimone deve firmare e datare personalmente la dichiarazione di consenso informato dopo che il modulo stesso e qualsiasi altra informazione scritta siano stati letti e spiegati al soggetto e questi abbia espresso il consenso verbale alla partecipazione allo studio.

### 78. Informativa e manifestazione del consenso al trattamento dei dati personali (1)

79. (Ai sensi delle linee guida per i trattamenti di dati personali nell'ambito delle sperimentazioni cliniche di medicinali - 24 luglio 2008 **G.U. n. 190 del 14 agosto 2008** e in conformità con il Testo unico D.L. 30 giugno 2003 n. 196 "Codice in materia di protezione dei dati personali")

80.

# 81. IL GARANTE PER LA PROTEZIONE DEI DATI PERSONALI

82.

#### 83. Titolari del trattamento e relative finalità

- 84. Il Promotore U.O. Ematologia degli Spedali Civili di Brescia, che ha commissionato lo studio che Le è stato descritto, in accordo alle responsabilità previste dalle norme della buona pratica clinica (d.l. 211/2003), tratterà i Suoi dati personali, in particolare quelli sulla salute, soltanto nella misura in cui sono indispensabili in relazione all'obiettivo dello studio.
- 85. A tal fine i dati indicati saranno raccolti e conservati dal Promotore.
- 86. Il trattamento dei dati personali relativi al suo stato di salute è indispensabile allo svolgimento dello studio: il rifiuto di conferirli non Le consentirà di parteciparvi.

#### 87. Natura dei dati

88. Il medico che La seguirà nello studio La identificherà con un codice: i dati che La riguardano raccolti nel corso dello studio, ad eccezione del Suo nominativo, saranno conservati dal Promotore, registrati, elaborati e unitamente a tale codice, alla Sua data di nascita, al sesso, al Suo peso e alla Sua statura. Soltanto il medico e i soggetti autorizzati potranno collegare questo codice al Suo nominativo.

89.

## 90. Modalità del trattamento

91. I dati, trattati mediante strumenti anche elettronici, saranno diffusi solo in forma rigorosamente anonima, ad esempio attraverso pubblicazioni scientifiche, statistiche e convegni scientifici. La Sua partecipazione allo studio implica che, in conformità alla normativa sulle sperimentazioni cliniche dei medicinali, il personale del Promotore, il Comitato etico e le autorità sanitarie italiane potranno conoscere i dati che La riguardano, contenuti anche nella Sua documentazione clinica originale, con modalità tali da garantire la riservatezza della Sua identità.

#### 92. Esercizio dei diritti

**93.** Potrà esercitare i diritti di cui all'art. 7 del Codice (es. accedere ai Suoi dati personali, integrarli, aggiornarli, rettificarli, opporsi al loro trattamento per motivi legittimi, ecc.) rivolgendosi direttamente al Promotore. Potrà interrompere in ogni momento e senza fornire alcuna giustificazione la Sua partecipazione allo studio: in tal caso, i dati a Lei correlati verranno distrutti.

Non saranno inoltre raccolti ulteriori dati che La riguardano, ferma restando l'utilizzazione di quelli eventualmente già raccolti per determinare, senza alterarli, i risultati della ricerca.

# 94.

# 95. Consenso

Sottoscrivendo tale modulo acconsento al trattamento dei miei dati personali per gli scopi della ricerca nei limiti e con le modalità indicate nell'informativa fornitami con il presente documento.

| 96. |
|---|
| 97. Nome e Cognome dell'interessato (in stampatello) |
| 98. Firma dell'interessato |
| 99. <b>Data</b> |
| 100. |
| 101. |
| 102. (1) Da sottoporre agli interessati unitamente al modulo di consenso informato che descrive |
| le caratteristiche scientifiche dello studio, anche mediante integrazione dello stesso. |
| 103. |
| 104. |